CLINICAL TRIAL: NCT05933694
Title: A Randomized Controlled Trial Comparing Performance of Primary Care Clinicians in the Interpretation of SPIROmetry With or Without Artificial Intelligence Decision Support Software
Brief Title: Spirometry Interpretation Performance of Primary Care Clinicians With/Without AI Software
Acronym: SPIRO-AID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 323361
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Lung Disease
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants to report 50 spirometry records alone
- Intervention (Experimental): Participants report the same 50 spirometry records provided in the control arm with an artificial intelligence-powered spirometry interpretation report
  Interventions: Other: Artificial Intelligence-powered Spirometry Interpretation Report

INTERVENTIONS:
Other: Artificial Intelligence-powered Spirometry Interpretation Report — A report generated by artificial intelligence powered software that assessed technical quality of spirometry and estimates the diagnostic probability of six categories: COPD/Asthma/ILD/ Normal/Other obstructive/Other Unidentified
  Other Names: ArtiQ.Spiro
  Arms: Intervention

SUMMARY:
To evaluate whether an artificial intelligence decision support software (ArtiQ.Spiro) improves the diagnostic accuracy of spirometry interpreted by primary care clinicians, as measured by Clinician Diagnostic Accuracy (vs Reference Standard).

DETAILED DESCRIPTION:
This is a randomised controlled study to evaluate the effects of AI support software on the performance of primary care clinicians in the interpretation of spirometry. Clinicians will be provided with a clinical dataset of 50 entirely anonymous, previously recorded real-world spirometry records to interpret and will be asked to complete specific questions about diagnosis and quality assessment. The records will be randomly selected from a database comprising spirometry records from 1122 patients undergoing spirometry in primary care and community -based respiratory clinics in Hillingdon borough between 2015-2018.

Participating clinicians will be allocated at random to receive either spirometry records alone or spirometry records with the addition of an AI spirometry interpretation eport. The clinical spirometry records will be de-identified (name, date of birth, address, postcode, occupation, GP, medications data removed), by a member of the clinical care team.

Study participants (participating clinicians) will independently examine the same 50 spirometry records through an online platform. For each spirometry record, the primary care clinician participant will answer questions about technical quality, pattern interpretation, preferred diagnosis, differential diagnosis and self-rated confidence with these answers.

The study statistician will be blinded to treatment allocation up to completion of analysis and interpretation.

The reference standards for spirometry technical quality and pattern interpretation will be made by a senior experienced respiratory physiologist but without access to AI report.

The reference standard for diagnosis will be made by a panel of three respiratory specialists from the clinical care team with access to medical notes and results of relevant investigations but without access to AI report.

ELIGIBILITY:
Inclusion Criteria:

1. Clinicians working in primary care (for at least 50% of their job plan) in the UK, who refer for or perform spirometry (typically GP, practice nurse)
2. Able to access spirometry traces on study platform
3. Provide written informed consent via study platform

Exclusion Criteria:

1. Clinicians who have completed specialist training in respiratory medicine and recognised by the General Medical Council with a right to practise as a NHS consultant in respiratory medicine

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2024-06-27 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Preferred Diagnostic Performance | Six months
  A correct case is where the preferred diagnosis matches the reference final diagnosis. Units will be percentage of total cases that are correct.

SECONDARY OUTCOMES:
Pattern interpretation | Six months
  A correct case is where the participants' selected pattern matches the reference pattern. Options are: Normal, Airflow obstruction, Possible restriction or non-specific pattern, Possible Mixed Disorder. Units will be percentage of total cases that are correct.
Differential diagnostic performance | Six months
  A correct case is where the preferred or differential diagnosis matches the reference final diagnosis. Units will be percentage of total cases that are correct.
Quality assessment performance | Six months
  A correct case is where the participant's quality grade matches the reference quality grade. Options are: Acceptable (Grade A/B) or Not Acceptable (Grades C/D/E/F/U). Units will be percentage of total cases that are correct.
Pattern interpretation self-rated confidence | Six months
  Pattern interpretation self-rated confidence will be measured on a visual analogue scale (0-10) where 0 = not confident at all; 10= very confident)
Diagnostic self-rated confidence | Six months
  Diagnostic self-rated confidence will be measured on a visual analogue scale (0-10) where 0 = not confident at all; 10= very confident)
Quality Assessment self-rated confidence | Six months
  Quality Assessment self-rated confidence will be measured on a visual analogue scale (0-10) where is 0 = not confident at all; 10= very confident)

CONTACTS AND LOCATIONS:
Overall Officials: William Man, Principal Investigator — Royal Brompton & Harefield Hospitals
Locations (1):
- Royal Brompton & Harefield Hospitals, Uxbridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Doe G, El-Emir E, Edwards GD, Topalovic M, Evans RA, Russell R, Sylvester KP, Van Orshoven K, Sunjaya AP, Scott DA, Prevost AT, Harvey J, Taylor SJ, Hopkinson NS, Kon SS, Jarrold I, Spain N, Banya W, Man WD. Comparing performance of primary care clinicians in the interpretation of SPIROmetry with or without Artificial Intelligence Decision support software (SPIRO-AID): a protocol for a randomised controlled trial. BMJ Open. 2024 Jul 1;14(6):e086736. doi: 10.1136/bmjopen-2024-086736. PMID 38950987